CLINICAL TRIAL: NCT05078788
Title: Efficacy of Holmium Laser Uretherotomy in Combination With Intralesional Steroids in the Treatment of Bulbar Uretheral Stricture
Brief Title: Holmium Laser Uretherotomy in Combination With Intralesional Steroids in Bulbar Uretheral Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M D 98/ 2020
Record Dates: First submitted 2021-09-21; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser uretherotomy (Experimental): Using Holmium laser uretherotomy only in the treatment of bulbar uretheral stricture
  Interventions: Procedure: Laser uretherotomy
- Laser uretherotomy with intralesional steroids (Experimental): Using holmium laser uretherotomy with injection of 80 mg of triamcinolone (diluted with normal saline to 10 ml) in the treatment of bulbar uretheral stricture
  Interventions: Procedure: Laser uretherotomy with triamcinolone

INTERVENTIONS:
Procedure: Laser uretherotomy — Holmium YAG Laser with pulse energy from 1-2 Joule, frequency from 10-15 Hertz and total power from 3.0 to 30.0 Watt were set up, respectively, based on the extent of the lesions. Scar tissue was incised at the position of 12-o'clock under the guidance of guidewire or ureteric catheter till fresh mucosa appeared.
  Arms: Laser uretherotomy
Procedure: Laser uretherotomy with triamcinolone — After laser urethrotomy, 80 mg of triamcinolone (diluted with normal saline to 10 ml) will be injected by using an injection needle (5 F size and 23 G needle size) at 10 sites, 1 ml each, along the site of urethrotomy and circumferentially.
  Arms: Laser uretherotomy with intralesional steroids

SUMMARY:
the purpose is to evaluate the outcome of visual internal uretherotomy with Holmium laser along with intralesional steroid injection.

DETAILED DESCRIPTION:
In this study, the investigator evaluates the efficacy of Holmium laser in combination with intra lesional steroid injection in the treatment of bulbar urethral strictures

ELIGIBILITY:
Inclusion Criteria:

1. Presence of obstructive symptoms,
2. Short segment strictures (stricture length <2 cm) as evident on radiological studies, i.e. retrograde urethrography and micturating cystourethrography.
3. Peak flow rate on uroflowmetry less than 15 ml/s

Exclusion Criteria:

1. Complete obliteration of lumen of urethra on urethroscopy,
2. Balanitis Xerotica Obliterans,
3. Age less than 18 years,
4. Multiple strictures,
5. Active urinary tract infection,
6. Recurrent Strictures.
7. Prior internal uretherotomy
8. Prior urethroplasty
9. Pan-anterior urethral strictures
10. Posterior stenosis
11. Those who lost to follow up

Ages: 26 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
the maximum flow rate (Qmax) is >15 ml/s at 3 and 6 months after procedure | 3 and 6 months
  The procedure will be accepted as successful when the maximum flow rate (Qmax) is >15 ml/s.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt